CLINICAL TRIAL: NCT03363165
Title: Hepatocyte Growth Factor to Improve Functioning in Peripheral Artery Disease: The HI-PAD Study
Brief Title: Hepatocyte Growth Factor to Improve Functioning in PAD
Acronym: HI-PAD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Helixmith Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Mary McDermott, Professor of Medicine at Northwestern University Feinberg School of Medicine, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU00205511; R21AG056903 (NIH)
Record Dates: First submitted 2017-11-30; First posted 2017-12-06 (Actual); Results first posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Peripheral Artery Disease
Keywords: PAD
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VM202 (Active Comparator): Participants will receive injections of VM202 (4 mgs) in calf skeletal muscle every 14 days for a total of four treatment days.
  Interventions: Drug: VM202
- Placebo (Placebo Comparator): Participants will receive injections of placebo in calf skeletal muscle every 14 days for a total of four treatment days.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: VM202 — Participants randomized to VM202 will receive calf muscle injections of VM202 to each leg with evidence of PAD. Injections of VM202 are administered by a physician in a double-blinded fashion after randomization on Day 0, Day 14, Day 28, and Day 42, for a total of four treatment days. Therefore, participants randomized to VM202 will receive 4 mgs of VM202 in each calf muscle on each treatment day. Injections are placed beginning 2 cm below the popliteal crease, and are administered in a pre-designed sequence and pattern, at a measured distance 2 cm apart.
  Note: Participants who have a evidence of PAD in only one leg will only receive injections in the leg with evidence of PAD.
  Arms: VM202
Other: Placebo — Participants randomized to placebo will receive calf muscle injections of placebo (the excipient buffer formulation minus the VM202) to each leg with evidence of PAD. Injections of placebo are administered by a physician in a double-blinded fashion after randomization on Day 0, Day 14, Day 28, and Day 42, for a total of four treatment days. Placebo appears identical to the VM202 study drug and is administered in a pattern on the calf identical to that of the VM202 injections.
  Note: Participants who have a evidence of PAD in only one leg will only receive injections in the leg with evidence of PAD.
  Arms: Placebo

SUMMARY:
HI-PAD is a placebo controlled double-blind randomized pilot clinical trial to determine whether VM202 may improve walking ability in people with lower extremity peripheral artery disease (PAD).

DETAILED DESCRIPTION:
The HI-PAD study will randomize 39 people age 55 and older with PAD who do not have critical limb ischemia. The primary outcome is change in the six-minute walk distance at 6-month follow-up after the first study drug injection. A secondary outcome in change in six-minute walk distance at 3-month follow-up. Additional secondary outcomes are pain-free and maximal treadmill walking distance, calf biopsy measures of skeletal muscle regeneration, capillary density, and autophagy, and MRI-measured calf muscle perfusion at three-month follow-up. Investigators will also measure change in six-minute walk distance at 12-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age 55 or above
* Symptomatic PAD, defined as exertion-induced ischemic calf muscle symptoms during the six-minute walk, during the baseline exercise stress test, or during daily walking activities. PAD will be defined as an ankle brachial index (ABI) < or = 0.90 at the baseline study visit or vascular lab evidence of PAD or angiographic evidence of significant PAD.

Exclusion Criteria:

* Above- or below-knee amputation.
* Critical limb ischemia, including individuals with gangrene and lower extremity ulcers.
* Wheelchair-bound or requiring a cane or walker to ambulate.
* Walking is limited by a symptom other than PAD.
* Lower extremity revascularization, orthopedic surgery, cardiovascular event, coronary revascularization, or other major surgery in the previous three months and planned revascularization or major surgery during the next six months.
* Major medical illness including renal disease requiring dialysis, lung disease requiring oxygen, Parkinson's disease, or a life-threatening illness with life expectancy less than six months. [NOTE: Participants who only use oxygen at night may still qualify]
* History of cancer within the last 5 years or incomplete cancer screening as recommended by the American Cancer Society. Specifically, participants will be asked to provide documentation regarding screening history for colon cancer and breast and cervical cancer (women), according to the American Cancer Society guidelines. Screening for colon cancer may consist of stool testing for blood in the past year. Men must either provide documentation regarding prostate cancer screening history or indicate after a telephone or in-person discussion with Dr. McDermott that they have elected to decline prostate cancer screening. A chest computed tomography will be performed for participants 55 to 74 years old with >30 pack year history of smoking, unless they have not smoked within the past 15 years, to screen for lung cancer that may exclude them. The study team may also perform colon, breast, and/or cervical cancer screenings as part of study participation. The study team will provide stool testing for blood for colon cancer screening, mammogram for breast cancer screening, and a Pap test for cervical cancer screening according to the participant's eligibility for these screening tests, using the American Cancer Society guidelines. Men who elect to have prostate cancer screening who have not had this completed with their physician can have a prostate specific antigen (PSA) test performed by study investigators. Participants who have a history of non-melanoma skin cancer (i.e.had basal cell carcinoma or squamous cell carcinoma of the skin) may still be eligible if the lesion was completely removed and there has been no evidence of recurrence in the past year.
* Evidence of proliferative retinopathy. Participants who were treated for retinopathy at least 5 years prior to their baseline assessment who do not have evidence of proliferative retinopathy at the time of baseline assessment may still be eligible.
* Positive test for active Human Immunodeficiency Virus (HIV), hepatitis B virus, hepatitis C virus or Human T-lymphotropic virus. Patients who have positive antibodies for HIV, hepatitis B, or hepatitis C who do not have detectable viral load will be eligible for participation.
* Mini-Mental Status Examination (MMSE) score <23 or dementia.
* Participation in or completion of a clinical trial in the previous three months. [NOTE: after completing a stem cell or gene therapy intervention, participants will become eligible after the final study follow-up visit of the stem cell or gene therapy study so long as at least six months have passed since the final intervention administration. After completing a supplement or drug therapy (other than stem cell or gene therapy), participants will be eligible after the final study follow-up visit as long as at least three months have passed since the final intervention of the trial.]
* Increase in angina or angina at rest.
* Premenopausal women.
* Non-English speaking.
* Visual impairment that limits walking ability.
* In addition to the above criteria, investigator discretion will be used to determine if the trial is unsafe or not a good fit for the potential participant.
* Potential participants who have had symptoms from peripheral artery disease for less than six months will be excluded.
* Potential participants who, after being advised of therapeutic options available for people with PAD, prefer to return to their physician to discuss alternative treatment (e.g. supervised exercise or revascularization). Potential participants may participate in the study after 12 weeks has passed since their last supervised exercise session or revascularization if they meet inclusion criteria.
* Potential participants with a baseline six-minute walk value < 595 or > 1,520 feet will be excluded.
* Potential participants with the following laboratory values will be excluded: a hemoglobin value < 8.0 g/dL, a white blood cell count < 3,000 cells per microliter, platelet count < 75,000/mm3, GFR < 20 mL/minute/1.73 M2, AST or ALT value > 3 times the upper limit of normal, or any other clinically significant laboratory abnormality which, in the opinion of the investigator, should exclude the participant. Participants may undergo a serum electrophoresis and an immunofixation blood test if indicated to further evaluate abnormalities on the complete blood count if needed to assess study eligibility.
* Potential participants started on cilostazol within the past three months will be excluded. They may be evaluated for eligibility once three months has passed since beginning cilostazol.
* Vulnerable populations (fetuses, pregnant women, children, prisoners, and institutionalized persons) and adults unable to consent will not be included in the study.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2023-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary McDermott, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nayak P, Polonsky T, Tian L, Greenland P, Xu S, Zhang D, Zhao L, Criqui MH, Kibbe MR, Gladders B, Goodney P, Ho K, Guralnik JM, McDermott MM. Medical therapies, comorbid conditions, and functional performance in people with peripheral artery disease enrolled in clinical trials between 2004 and 2021. Vasc Med. 2023 Apr;28(2):144-146. doi: 10.1177/1358863X221145533. Epub 2023 Jan 1. PMID 36588397

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants will receive injections of placebo in calf skeletal muscle every 14 days for a total of four treatment days.
  Placebo: Participants randomized to placebo will receive calf muscle injections of placebo (the excipient buffer formulation minus the VM202) to each leg with evidence of PAD. Injections of placebo are administered by a physician in a double-blinded fashion after randomization on Day 0, Day 14, Day 28, and Day 42, for a total of four treatment days. Placebo appears identical to the VM202 study drug and is administered in a pattern on the calf identical to that of the VM202 injections.
  Note: Participants who have a evidence of PAD in only one leg will only receive injections in the leg with evidence of PAD.
- VM202: Participants will receive injections of VM202 (4 mgs) in calf skeletal muscle every 14 days for a total of four treatment days.
  VM202: Participants randomized to VM202 will receive calf muscle injections of VM202 to each leg with evidence of PAD. Injections of VM202 are administered by a physician in a double-blinded fashion after randomization on Day 0, Day 14, Day 28, and Day 42, for a total of four treatment days. Therefore, participants randomized to VM202 will receive 4 mgs of VM202 in each calf muscle on each treatment day. Injections are placed beginning 2 cm below the popliteal crease, and are administered in a pre-designed sequence and pattern, at a measured distance 2 cm apart.
  Note: Participants who have a evidence of PAD in only one leg will only receive injections in the leg with evidence of PAD.
Period: 3-month Follow-up
Arm/Group | Placebo | VM202
Started | 18 | 21
Completed | 18 | 20
Not Completed | 0 | 1
Not completed — Death | 0 | 1
Period: 6-month Follow-up
Arm/Group | Placebo | VM202
Started | 18 | 21
Completed | 17 | 19
Not Completed | 1 | 2
Not completed — Death | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1
Period: 12-month Follow-up
Arm/Group | Placebo | VM202
Started | 18 | 21
Completed | 16 | 19
Not Completed | 2 | 2
Not completed — Death | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VM202 | Placebo | Total
Number analyzed (Participants) | 21 | 18 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.9 (8.9) | 67.1 (7.0) | 69.1 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 14 | 14 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 20 | 18 | 38
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 10 | 25
  White | 5 | 7 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Ankle Brachial Index [Mean (Standard Deviation); unit: ratio of systolic pressures] — A ratio of Doppler recorded systolic pressures in the lower and upper extremity arteries.
  ratio of systolic pressures | 0.61 (0.12) | 0.63 (0.13) | 0.62 (0.12)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 29.8 (6.4) | 30.0 (5.6) | 29.9 (6.0)
Six-minute walk distance [Mean (Standard Deviation); unit: meters] | 321.7 (72.2) | 310.2 (77.9) | 316.4 (74.1)

OUTCOME MEASURES:

1. Primary Outcome: Six-minute Walk Distance
Description: Participants walking up and down a 100 foot hallway for six minutes following a standardized protocol. The goal is for them to walk as far as possible in six minutes
Time Frame: Change from baseline to six-month follow-up in six-minute walk distance
Measure: Mean (Standard Error); unit: meters
Arm/Group | Placebo | VM202
Number analyzed (Participants) | 17 | 19
meters | 17.01 (13.76) | 3.46 (12.70)
Statistical Analysis 1: Comparison: Placebo vs VM202; Test type: Superiority; p = 0.7586, ANCOVA; Adjusted for baseline six-minute walk distance, age, race, former smoker; Mean Difference (Final Values) = -13.54, 90% CI 1-sided [lower limit -38.52]

2. Secondary Outcome: Maximal Treadmill Walking Time
Description: A Gardner or Modified Gardner treadmill exercise protocol will be used
Time Frame: Change from baseline to three-month follow-up
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Placebo | VM202
Number analyzed (Participants) | 8 | 10
minutes | -0.59 (0.73) | 1.66 (0.73)
Statistical Analysis 1: Comparison: Placebo vs VM202; Test type: Superiority; p = 0.0298, ANCOVA; Adjusted for baseline maximal treadmill walking time, age, race, former smoker; Mean Difference (Final Values) = 2.25, 90% CI 1-sided [lower limit 0.78]

3. Secondary Outcome: Calf Muscle Perfusion
Description: Calf muscle perfusion is measured by Magnetic Resonance Imaging (MRI) Unit of measure is ml/minute per 100 gms tissue
Time Frame: Change from baseline to three-month follow-up
Measure: Mean (Standard Error); unit: ml/minute per 100 gm tissue
Arm/Group | Placebo | VM202
Number analyzed (Participants) | 6 | 7
ml/minute per 100 gm tissue | 1.98 (1.90) | 2.68 (1.87)
Statistical Analysis 1: Comparison: Placebo vs VM202; Test type: Superiority; p = 0.4019, ANCOVA; Adjusted for baseline perfusion, age, race, former smoker; Mean Difference (Final Values) = 0.69, 90% CI 1-sided [lower limit -3.10]

4. Secondary Outcome: Calf Muscle Biopsy Biochemical Measures (Satellite Cells - Total SCs/100 Fibers)
Description: A skeletal muscle sample will be obtained from the calf muscle. The outcome is the number of satellite cells per 100 muscle fibers
Time Frame: Change from baseline to three-month follow-up
Measure: Mean (Standard Error); unit: Satellite cells per 100 muscle fibers
Arm/Group | Placebo | VM202
Number analyzed (Participants) | 5 | 7
Satellite cells per 100 muscle fibers | -4.83 (8.23) | 3.45 (6.91)
Statistical Analysis 1: Comparison: Placebo vs VM202; Test type: Superiority; p = 0.2080, ANCOVA; Adjusted for baseline muscle measure, age, race, former smoker; Mean Difference (Final Values) = 8.28, 90% CI 1-sided [lower limit -5.37]

5. Secondary Outcome: Walking Impairment Questionnaire - Distance Score
Description: The well validated Walking Impairment Questionnaire will be used to measure patient- perceived walking performance. The WIQ is scored from 0-100, with 100 being the best score. We will use distance and speed sub-components separately.
Time Frame: Change from baseline to three-month follow-up
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | VM202
Number analyzed (Participants) | 17 | 20
score on a scale | 6.28 (5.54) | 8.30 (5.19)
Statistical Analysis 1: Comparison: Placebo vs VM202; Test type: Superiority; p = 0.3980, ANCOVA; Adjusted for baseline WIQ distance score, age, race, former smoker; Mean Difference (Final Values) = 2.02, 90% CI 1-sided [lower limit -8.11]

6. Secondary Outcome: The Short-Form-36 Physical Functioning Score
Description: This well validated quality of life measure will be used to assess changes in patient perceived quality of life. The SF-36 is scored from 0-100, with 100 being the best score.
Time Frame: Change from baseline to three-month follow-up
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | VM202
Number analyzed (Participants) | 17 | 20
score on a scale | 8.70 (4.94) | 3.20 (4.60)
Statistical Analysis 1: Comparison: Placebo vs VM202; Test type: Superiority; p = 0.7852, ANCOVA; Adjusted for baseline SF-36 physical functioning score, age, race, former smoker; Mean Difference (Final Values) = -5.50, 90% CI 1-sided [lower limit -14.50]

7. Secondary Outcome: The Short-Form-36 Physical Functioning Score
Description: This well validated quality of life measure will be used to assess changes in patient perceived quality of life. Scored on a 0-100 scale, where 100- is best.
Time Frame: Change from baseline to six-month follow-up
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | VM202
Number analyzed (Participants) | 17 | 20
score on a scale | 11.98 (3.67) | 6.84 (3.32)
Statistical Analysis 1: Comparison: Placebo vs VM202; Test type: Superiority; p = 0.8414, ANCOVA; Adjusted for baseline SF-36 physical functioning score, age, race, former smoker; Mean Difference (Final Values) = -5.14, 90% CI 1-sided [lower limit -11.76]

8. Secondary Outcome: Walking Impairment Questionnaire - Distance Score
Description: The well validated Walking Impairment Questionnaire will be used to measure patient- perceived walking performance.
Time Frame: Change from baseline to six-month follow-up
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | VM202
Number analyzed (Participants) | 17 | 20
score on a scale | 11.44 (6.63) | 9.31 (6.01)
Statistical Analysis 1: Comparison: Placebo vs VM202; Test type: Superiority; p = 0.5912, ANCOVA; Adjusted for baseline WIQ distance score, age, race, former smoker; Mean Difference (Final Values) = -2.13, 90% CI 1-sided [lower limit -14.11]

9. Secondary Outcome: Six-minute Walk Distance
Description: as for outcome 1
Time Frame: Change in six-minute walk distance from baseline to three-month follow-up
Measure: Mean (Standard Error); unit: meters
Arm/Group | Placebo | VM202
Number analyzed (Participants) | 17 | 20
meters | -0.48 (12.80) | -2.49 (12.01)
Statistical Analysis 1: Comparison: Placebo vs VM202; Test type: Superiority; p = 0.5442, ANCOVA; Adjusted for baseline six-minute walk distance, age, race, former smoker; Mean Difference (Final Values) = -2.00, 90% CI 1-sided [lower limit -25.47]

10. Secondary Outcome: Pain-free Treadmill Walking Time
Description: A Gardner or Modified Gardner treadmill exercise protocol will be used
Time Frame: Change from baseline to three-month follow-up
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Placebo | VM202
Number analyzed (Participants) | 8 | 10
minutes | 0.95 (0.80) | 0.45 (0.77)
Statistical Analysis 1: Comparison: Placebo vs VM202; Test type: Superiority; p = 0.6603, ANCOVA — Adjusted for baseline pain-free treadmill walking time, age, race, former smoker; Mean Difference (Final Values) = -0.50, 90% CI 1-sided [lower limit -2.11]

11. Other Pre Specified Outcome: Six-minute Walk Distance
Description: See above regarding 6-minute walk protocol
Time Frame: Change from baseline to 12-month follow-up in six minute walk distance.
Measure: Mean (Standard Error); unit: meters
Arm/Group | Placebo | VM202
Number analyzed (Participants) | 16 | 18
meters | 5.02 (12.17) | 2.24 (11.17)
Statistical Analysis 1: Comparison: Placebo vs VM202; Test type: Superiority; p = 0.5647, ANCOVA; Adjusted for baseline six-minute walk distance, age, race, former smoker; Mean Difference (Final Values) = -2.78, 90% CI 1-sided [lower limit -24.99]

ADVERSE EVENTS:
Time Frame: Adverse events forms are collected at 2nd, 3rd, and 4th injection days, as well as the 3-month, 6-month, and 12-month follow-up visits.
Arm/Group | Placebo | VM202
All-Cause Mortality (participants affected / at risk) | 1/18 | 1/21
Serious Adverse Events (participants affected / at risk) | 6/18 | 6/21
Other Adverse Events (participants affected / at risk) | 14/18 | 17/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=18) | VM202 (N=21)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 0 (0)
Lower extremity revascularization (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Fall and fracture (General disorders) | 0 (0) | 1 (1)
Dehydration (General disorders) | 1 (1) | 0 (0)
Bowel obstruction (General disorders) | 1 (1) | 0 (0)
Colonoscopy (General disorders) | 1 (1) | 0 (0)
Palpitations and anemia (General disorders) | 0 (0) | 1 (1)
Blood transfusion/anemia (General disorders) | 0 (0) | 1 (1)
COVID-19 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulled muscle (General disorders) | 0 (0) | 1 (1)
Hypertension (General disorders) | 0 (0) | 1 (1)
COPD exacerbation (General disorders) | 1 (1) | 0 (0)
Lower extremity arterial bypass surgery (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=18) | VM202 (N=21)
Pain or discomfort at the study drug injection sites (General disorders) | 7 (8) | 13 (24)
Redness or irritation at the study drug injection sites (General disorders) | 3 (3) | 4 (6)
Diagnosed with infection at any of the injection sites (General disorders) | 0 (0) | 0 (0)
Venous thromboembolism (deep venous thrombosis or pulmonary embolism) (General disorders) | 0 (0) | 2 (2)
Eye disease - proliferative retinopathy (General disorders) | 0 (0) | 0 (0)
Diagnosed with a new tumor or cancer (General disorders) | 0 (0) | 0 (0)
Stayed overnight in the hospital (General disorders) | 6 (8) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-12): https://cdn.clinicaltrials.gov/large-docs/65/NCT03363165/Prot_SAP_001.pdf